CLINICAL TRIAL: NCT06807047
Title: The Effect of Epilepsy Management at School Mobile Health Application on Epilepsy Knowledge, Attitudes, and Self-Management of Teachers of Children With Intellectual Disability: A Randomized Controlled Study
Brief Title: Effect of the EpiSchool-M App on Teachers' Epilepsy Knowledge, Attitudes, and Self-Management
Acronym: EpiSchool-M
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafkas University (Other)
Collaborators: Akdeniz University (Other)
Responsible Party: Principal Investigator, Zahide İYİ ALTINIŞIK, Resarch Assistant, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KAEK-33
Record Dates: First submitted 2025-01-23; First posted 2025-02-04 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Epilepsy; Intellectual Disabilities; Teacher Training; Mobile Applications; Knowledge; Attitude; Self Management
Keywords: epilepsy; children with intellectual disabilities; Mobile Health Application; epilepsy knowledge; epilepsy attitude; epilepsy self management
MeSH Terms: conditions — Epilepsy; Intellectual Disability; Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Mobile Application Group (Experimental): Teachers in the Epilepsy Management at School Mobile Health Application group will download the EpiSchool app to their phones. Within two weeks, they will watch the epilepsy-related educational videos and the animation video integrated into the app.
  Interventions: Other: Epilepsy Management at School Mobile Health Application
- Digital Education Guide Group (Experimental): The digital guide, prepared based on expert opinions, will be sent to the teachers via a link. They will be asked to read the guide within 15 days.
  Interventions: Other: Digital Epilepsy Education Guide
- Control Group (No Intervention): Group without any intervention

INTERVENTIONS:
Other: Epilepsy Management at School Mobile Health Application — Teachers who meet the inclusion criteria will use the EpiSchool
  Arms: Mobile Application Group
Other: Digital Epilepsy Education Guide — Teachers who meet the inclusion criteria will use the EpiGuide
  Arms: Digital Education Guide Group

SUMMARY:
The aim of this study was to determine the effects of the training given to the teachers of children with intellectual disabilities with the "Epilepsy Management at School Mobile Health Application" and the "Digital Epilepsy Education Guide" on teachers' epilepsy knowledge, attitudes, and self management levels. This study was planned in a pretest, posttest design, follow-up, randomized controlled study. The sample of the study will consist of 90 teachers. Intervention-1 (Epilepsy Management at School Mobile Health Application, n=30), intervention-2 (Digital Epilepsy Education Guide, n=30) and control group (group without any intervention, n=30) will be included in the study. The data collection tools to be used in the research will be applied to all three groups at the same time intervals (T0: Just before the application phase of the research, T1: 15 days after the application, T2: one month after the application). The data will be collected using the Personal Information Form, the Knowledge and Attitudes Toward Epilepsy Among School Teachers Scale, and the Epilepsy Self-Management Scale for Teachers. Statistical Package for the Social Sciences (SPSS) 25.0 package program will be used in the analysis of the data.

ELIGIBILITY:
Inclusion Criteria:

* Working at special education schools affiliated with the Ministry of National Education in Antalya Province,
* Teachers of children with moderate to severe intellectual disabilities,
* Having a smartphone with internet access and either an Android or iOS operating system.

Exclusion Criteria:

* Teachers of children with hearing and visual impairments, without intellectual disabilities
* Teachers of children with mild intellectual disabilities

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2025-03-10 (Actual); Primary Completion 2025-03-24 (Actual); Study Completion 2025-04-24 (Actual)

PRIMARY OUTCOMES:
Knowledge And Attitudes Toward Epilepsy Among School Teachers Scale | 1.5 months
  The scales developed by Kos et al. (2023) assess knowledge and attitudes toward epilepsy. A higher total score indicates a higher level of knowledge and attitude. The scales consist of two parts: the "Attitudes Toward Epilepsy Among School Teachers Scale" and the "Knowledge Toward Epilepsy Among School Teachers Scale." The "Attitudes Toward Epilepsy Among School Teachers Scale" has two subdimensions: attitudes toward social relationships of children with epilepsy (10 items) and attitudes toward epilepsy-related limitations (5 items), totaling 15 items. A lower score on this scale indicates more positive attitudes toward epilepsy.
  The "Knowledge Toward Epilepsy Among School Teachers Scale" includes two subdimensions: knowledge about epilepsy (2 items) and knowledge about epilepsy's effects (10 items), totaling 12 items. A lower score on this scale indicates higher knowledge about epilepsy.
  Both scales are five-point Likert-type measurement tools.
Epilepsy Self-Management Scale for Teachers | 1.5 months
  The Epilepsy Self-Management Scale for Teachers, developed by Kos et al. (2022), aims to assess epilepsy self-management in teachers. It is a 23-item, five-point Likert scale. Responses are numbered from 1 to 5, with 1 meaning "Never" and 5 meaning "Always." Each item on the scale can receive a score between 1 and 5. The scale consists of three subdimensions: the first subdimension is seizure-related self-management (13 items), the second subdimension is pre-seizure self-management (5 items), and the third subdimension is post-seizure self-management (5 items).

CONTACTS AND LOCATIONS:
Locations (1):
- Akdeniz University, Antalya, Konyaaltı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided